CLINICAL TRIAL: NCT03753646
Title: Evaluating Effects of Integrating ECD Activities Into Bangladesh Government's Urban Lactating Mothers Allowance Program for the Poor on Children's Cognition and Behaviour in Rangpur City Corporation, Bangladesh
Brief Title: Evaluating Effects of Integrating ECD Activities Into Bangladesh Government's Urban Lactating Mothers Allowance Program for the Poor on Children's Cognition and Behavior in Rangpur City Corporation, Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR-18035
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Early Childhood Development
Keywords: Bangladesh; Cognitive development; behavior; quality of life; psycho social stimulation; lactating allowance
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: We will integrate ECD services to Bangladesh government lactating allowance to measure children's neurocognitive behavior in urban area of Bangladesh.
Who Masked: Outcomes Assessor
Masking Description: The Assessor who will measure children's cognitive development and behavor and other measurements will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactating allowance and psycho social stimulation (Experimental): Mothers will receive lactating allowance and psycho social stimulation
  Interventions: Other: Lactating allowance and psycho social stimulation
- Only lactating allowance (No Intervention): Mothers will receive only lactating allowance

INTERVENTIONS:
Other: Lactating allowance and psycho social stimulation — Mothers will receive lactating allowance and psycho social stimulation
  Arms: Lactating allowance and psycho social stimulation

SUMMARY:
Burden:

Provision of health care to urban poor population is a great challenge because of supply and demand barriers in the urban health system, which is considered patchy and fragmented. The poor urban people, especially mothers have little access to government health facilities. The health care platform is not well designed in primary health care delivery for urban health system but presently almost 30 percent people are living in urban area of the country.

Knowledge gap:

Little is known about what happen if psycho social stimulation is provided using urban lactating allowance program on children's cognition and behavior. There is little information about nature and bottleneck of Early Childhood Development (ECD) activities available in the urban Bangladesh.

Relevance:

This is an opportunity to develop a combined package integrating psycho social stimulation with the existing urban lactating allowance program on disadvantaged children's development.

As the urban health system is complex, patchy and fragmented, prior to this intervention An analysis will be done on ECD services and its bottleneck in urban area through Tanahashi framework.

Hypothesis (if any):

Adding psycho social stimulation to urban lactating allowance program will have additional effect on children's cognitive, motor and language development and behavior compared to the comparison group

Secondary Hypothesis:

Additionally the intervention will- improve mothers' quality of life and reduce their depressive symptoms be cost effective,

Objectives:

* To evaluate the effect of integrated urban lactating allowance and psycho social stimulation on children's cognitive, motor and language development and behavior
* To measure nature and bottleneck of ECD services in urban Bangladesh

Secondary objectives:

To measure effect of the programs on:

* mothers' quality of life and mental health (depression symptoms)
* cost effectiveness of the intervention

Methods: A two-arm, Cluster Randomized Controlled Trial: i) Lactating allowance + Psycho social stimulation; (ii) Only lactating allowance

Outcome measures/variables: Children's cognitive, motor and language development measured on Bayley-III, behavior on Wolke's rating scales, Mother's quality of life and depressive symptoms , household food security status, socioeconomic status, quality of home stimulation using family care indicators, Mother's knowledge on child care and development, children's growth measured by length/height, weight and head circumference,mothers' height, weight and mid upper arm circumference, direct and indirect cost of the project.

DETAILED DESCRIPTION:
It is estimated that 250 million children do not reach their potential due to poverty, inadequate stimulation and associated risk factors in low and middle income countries.

In Bangladesh more than 50% of children under 5 years are at risk of developmental delay. Urban population is about 28% and it is expected to rise to more than 40% by 2030. In fact, urbanization in Bangladesh is rapidly growing but is not well planned. Poor urban women and children are vulnerable in terms of health and education .

The urban health care facilities are fragmented and patchy and every year rise in population is putting more pressure on health system. Moreover, there is huge economic disparity between rich and poor in the urban areas and poorer people have little access to health care due to both supply and demand barriers. So the situation is rolling more difficult every day.

Ministry of Women and Children Affairs (MOWCA) has taken initiatives to help urban poor mothers through lactating allowance (LA) and limited health education programs. A study conducted in Zimbabwe documented that unconditional cash transfer showed an increase in receiving children's birth certificate and immunization in the age group of 0-4years and school attendance in 6-12 years. Recent systematic review concluded that unconditional cash transfer may not improve health services use in children and adult in low and middle income countries but may have positive impact on food choices and food security. It is expected that this urban lactating allowance will develop economic capacity of people, empower women, improve their quality of life and reduce gender gap.

Very few ECD programs are available for poor urban children especially for the 1st thousand days. The idea is to develop a combined package integrating psycho social stimulation with the existing urban lactating allowance program and measuring its effects on disadvantaged children's development.

As the urban health system is complex, patchy and fragmented, prior to this intervention an analysis will be done on ECD services and its bottleneck in the project area through Tanahashi framework. A facility assessment will be done to understand nature of ECD services. A meeting will be conducted with relevant experts to finalize the services delivery mechanism of the intervention.

Research Design and Methods:

This study will follow two sequential stages:

Stage I: Understand nature and analyse bottleneck of ECD services in selected urban areas of Bangladesh through a survey using Tanahasi framework.

Stage II: Document that adding ECD activities to urban lactating allowance program will improve children's cognition, motor, language and behaviour.

Methodology for stage I:

First, an analysis will be done on ECD program in urban area through Tanahashi framework. A documentation will be done on availability, accessibility, utilization and adequate coverage of the ECD activities.

ECD and related services will be analyzed through:

a) Household Survey and b) Facility assessment

1. Household survey A survey will be conducted with 426 mothers having child less than five years. On an average 22 respondents will be recruited from each cluster. the total clusters will be 20.

   Sample size was calculated assuming 50% effective coverage, 20% error, 95% confidence interval and 10% refusal rate the total sample size calculated was 426 in an urban setting..
2. Facility Assessment Moreover, ECD or relevant services will be collected through visiting service delivery facilities. government and private hospitals, NGOs and schools (kindergarten) will be visited and data will be collected on services available.

At the end of this stage, a stakeholders meeting with relevant experts will be conducted to finalize a service delivery mechanism

Methodology for stage II:

The main aim is to document that adding ECD activities to urban lactating allowance program improves children's cognition, language and motor and behaviour.

Study design:

This is a cluster randomized controlled trial of the effects of adding psycho social stimulation to the existing lactating allowance of the country with 2 arms: i) Psycho social stimulation+ Urban lactating allowance and ii) Only urban lactating allowance.

Selection of the study area:

A municipality will be selected for this study. The Initial plan is to conduct the study in Rangpur City Corporation.

Recruitment:

There will be 20 clusters (10 interventions & 10 comparisons) and 30 mother child dyads in each cluster. In Rangpure City Corporation there are 33 Wards. A Ward will be considered as a cluster. Cluster will be assigned randomly to intervention or comparisions group. A buffer zone will be made to reduce spill over effect with remaining Wards and or villages.

As the Government is providing urban lactating allowance to 2000 mothers in Rangpur City Corporation, it is expected that there will be approximately at least 50 mother child dyads in each cluster. 30 participants will be selected from the list considering mothers lower age and/or those with single child (if available).

Sample Size:

In total, sample is 600. Previous studies of psycho social stimulation alone achieved an effect size of 0.4 SD on children's development. In this study, lactating allowance (cash) as an intervention that might have also positive effect on the child development. But to be on the safe side, it is assumed that an effect size of 0.35 SD, 80% power, 95% confidence interval, 1.58 cluster design effect and 25% drop-out rate the sample size was calculated to be 300 in each arm with 30 children in each of the 20 clusters.

Data Analysis:

Data will be checked for normality. Appropriate measures will be taken if there are any abnormal distributions. Frequency table and percentage will be used to present nature of ECD services and its bottleneck. Service availability would be presented in a table through facility assessment and the bottlenecks (accessibility, utilization and coverage) will also be presented through interviews with mothers. For intervention trial, differences between groups in background characteristics will be analyzed using t-test for continuous variables and chi-square test for categorical variables.. Effect of the ECD intervention will be measured using intention-to-treat analysis controlling for the clustering effect in multivariate regression analysis. All covariates will be controlled and effect modifier and mulnicolinearity will be checked before regression analysis. Quality of life data will be analysed based on WHO guideline for WHOQoL tools.. Similarly, total score of SRQ will be calculated and then differences between arms will be analysed.

Cost-effectiveness Analysis:

The objective of the study is to estimate the resource use and costs associated with interventions. Direct and indirect cost will be measured for all the groups. Average costs per participants will be calculated by multiplying the cost of resource items by their respective unit costs. Outcomes will be generated from the study after the intervention and the differences will be measured before and after the intervention in two groups. Then the incremental cost-effectiveness ratio (ICER) will be used in cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a child aged 6-16 months
* Not expected to leave the study site for more than 2 months
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* Legal guardian unwilling or unable to provide written informed consent.
* Known congenital anomaly, developmental disorder or severe developmental delay
* If not possible to test the child due to physical or behavioural problems
* Children of multiple birth e.g. twin, triplets

Ages: 6 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Children's cognitive composite score ranging from 55 to 145 using Bayley Scales of Infant and Toddler Development (Bayley-III) | Children's cognitive composite score ranging from 55 to 145 using Bayley Scales of Infant and Toddler Development (Bayley-III) after one year intervention
  Children's cognitive composite score ranging from 55 to 145 using Bayley Scales of Infant and Toddler Development (Bayley-III). Higher values represent a better status
Children's language composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III) | Children's language composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III) after one year intervention
  Children's language composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III). Higher values represent a better status
Children's motor composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III) | Children's motor composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III) after one year intervention
  Children's motor composite score ranging from 45 to 155 using Bayley Scales of Infant and Toddler Development (Bayley-III). Higher values represent a better status
Children's approach behaviour using Wolk's behavior rating scale ranging from 1 to 9 | Children's approach behaviour using Wolk's behavior rating scale ranging from 1 to 9 after one year intervention
  Children's approach behaviour using Wolk's behavior rating scale ranging from 1 to 9 during Bayley. Higher values represent a better status
Children's general emotion tone behaviour using Wolk's behavior rating scale ranging from 1 to 9 | Children's general emotion tone behaviour using Wolk's behavior rating scale ranging from 1 to 9 after one year intervention
  Children's general emotion tone behaviour using Wolk's behavior rating scale ranging from 1 to 9 during Bayley. Higher values represent a better status
Children's activity behaviour using Wolk's behavior rating scale ranging from 1 to 9 | Children's activity behaviour using Wolk's behavior rating scale ranging from 1 to 9 after one year intervention
  Children's activity behaviour using Wolk's behavior rating scale ranging from 1 to 9 during Bayley. Higher values represent a more active status.
Children's cooperation behaviour using Wolk's behavior rating scale ranging from 1 to 9 | Children's cooperation behaviour using Wolk's behavior rating scale ranging from 1 to 9 after one year intervention
  Children's cooperation behaviour using Wolk's behavior rating scale ranging from 1 to 9 during Bayley. Higher values represent a better status
Children's vocalization behaviour using Wolk's behavior rating scale ranging from 1 to 9 | Children's vocalization behaviour using Wolk's behavior rating scale ranging from 1 to 9 after one year intervention
  Children's vocalization behaviour using Wolk's behavior rating scale ranging from 1 to 9 during Bayley. Higher values represent a better status

SECONDARY OUTCOMES:
Children's weight | Change children's weight after one year intervention
  Children's weight will be measured in Gram
Children's height | Change children's height after one year intervention
  Children's height will be measured in Gram
Children's Mid Upper Arm circumference (MUAC) | Change children's MUAC after one year intervention
  Children's MUAC will be measured by millimeter
Mothers' weight | Change mother's weight after one year intervention
  Mothers' weight will be measured in Gram
Mothers' height | Change mother's height after one year intervention
  Mothers' height will be measured by Centimeter
Mothers' Mid Upper Arm circumference (MUAC) | Change mother's Mid Upper Arm circumference (MUAC) after one year intervention
  Mothers' Mid Upper Arm circumference (MUAC) will be measured by Centimeter
Mothers' depressive symptom | Change mother's depression status after one year intervention
  Mothers' depressive symptom will be measured by Self-Regulation Questionnaire (SRQ). higher values represent a worse mental status
Mothers' quality of life status | Change mother's quality of life status after one year intervention
  Mothers' quality of life status will be measured by World Health Organization (WHO) quality of life questionnaire
Family's monthly food security status | Change family's food security status after one year intervention
  Family's monthly food security status will be measured by Household Food Insecurity Access Scale (HFIAS) questionnaire. The status will be measured as per HFIAS analysis guideline developed by the U.S. Agency for International Development (USAID).
  Measurement of Food Access:
  Indicator Guide
Domestic violence (mothers) | Change family's domestic violence status after one year intervention
  Domestic violence (mothers) monthly status will be measured by questionnaire
Family care indicators (FCI) | Change of FCI after one year intervention
  Family care indicators (FCI) will be measured by questionnaire. Higher values represent a better environment
Mothers' knowledge on parenting | Change of mothers' knowledge after one year intervention
  Mothers' knowledge on parenting questionnaire will be used

OTHER OUTCOMES:
Family's health seeking behavior | Change family's health seeking behaviour status after one year intervention
  Family's health seeking behavior status will be measured by questionnaire
Family's income | Change family's income status after one year intervention
  Family's monthly income status will be measured by questionnaire
Family's expenditure | Change family's expenditure status after one year intervention
  Family's expenditure status will be measured by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Background] Hamadani JD, Tofail F, Huda SN, Alam DS, Ridout DA, Attanasio O, Grantham-McGregor SM. Cognitive deficit and poverty in the first 5 years of childhood in Bangladesh. Pediatrics. 2014 Oct;134(4):e1001-8. doi: 10.1542/peds.2014-0694. PMID 25266433
- [Background] Afsana K, Wahid SS. Health care for poor people in the urban slums of Bangladesh. Lancet. 2013 Dec 21;382(9910):2049-51. doi: 10.1016/S0140-6736(13)62295-3. Epub 2013 Nov 21. No abstract available. PMID 24268606
- [Background] Robertson L, Mushati P, Eaton JW, Dumba L, Mavise G, Makoni J, Schumacher C, Crea T, Monasch R, Sherr L, Garnett GP, Nyamukapa C, Gregson S. Effects of unconditional and conditional cash transfers on child health and development in Zimbabwe: a cluster-randomised trial. Lancet. 2013 Apr 13;381(9874):1283-92. doi: 10.1016/S0140-6736(12)62168-0. Epub 2013 Feb 27. PMID 23453283
- [Background] Pega F, Liu SY, Walter S, Pabayo R, Saith R, Lhachimi SK. Unconditional cash transfers for reducing poverty and vulnerabilities: effect on use of health services and health outcomes in low- and middle-income countries. Cochrane Database Syst Rev. 2017 Nov 15;11(11):CD011135. doi: 10.1002/14651858.CD011135.pub2. PMID 29139110
- [Background] Ahmed SM, Evans TG, Standing H, Mahmud S. Harnessing pluralism for better health in Bangladesh. Lancet. 2013 Nov 23;382(9906):1746-55. doi: 10.1016/S0140-6736(13)62147-9. Epub 2013 Nov 21. PMID 24268003
- [Derived] Hossain SJ, Rahman SM, Fisher J, Rahman A, Tofail F, Hamadani JD. Effect of a parenting and nutrition education programme on development and growth of children using a social safety-net platform in urban Bangladesh: a cluster randomized controlled trial. Lancet Reg Health Southeast Asia. 2024 Mar 19;25:100388. doi: 10.1016/j.lansea.2024.100388. eCollection 2024 Jun. PMID 38550293